CLINICAL TRIAL: NCT00391885
Title: Target-controlled Infusion of Propofol and Remifentanil During General Anaesthesia Guided by Entropy of the Electroencephalogram: Comparison Between Manual Perfusion and Automated Perfusion
Brief Title: Target-controlled Infusion of Propofol and Remifentanil During General Anaesthesia Guided by Entropy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Foch-4
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Closed-loop anesthesia system

SUMMARY:
This study compares the manual administration of propofol and remifentanil and their delivery using a combined closed-loop anesthesia system, entropy of the EEG being the controller.

DETAILED DESCRIPTION:
Several monitors are currently proposed to evaluate the depth of hypnosis. Among them, Bispectral Index (BIS) is a well known and widely used parameter derived from the patient's electroencephalograph (EEG). A closed-loop anesthesia system can be built using BIS as the control variable, a proportional-integral-differential control algorithm, a propofol and a remifentanil target-controlled infusion systems as the control actuators Preliminary results show that this system can be used during surgery.

Spectral entropy relies on the extent of disorder in both EEG and electromyography (EMG) signals and returns 2 values: State Entropy (SE) and Response Entropy. SE is computed over the frequency range of 0.8-32 Hz and reflects the level of hypnosis while Response Entropy is computed over the frequency range of 0.8-47 Hz and reflects also EMG activity. BIS and SE are dimensionless numbers scaled from 100 to 0 for BIS and from 91 to 0 for SE. We hypothesized that SE can be used as the control variable. In preparation for a large multi-center control trial, we propose a prospective randomized study to evaluate the effectiveness of such a closed-loop anesthesia system. Two groups of patients are compared: one in which propofol and remifentanil are administered by the anesthesiologist using target-controlled infusion systems, and one in which propofol and remifentanil are administered automatically by the combined closed-loop anesthesia system. In both groups, the goal is to maintain SE between 40 and 60, the recommended range during anesthesia by the manufacturer. We expect the combined closed-loop anesthesia system group to do similar or better.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1-3,
* surgery under general anesthesia using relaxant agent,
* surgery lasting more than one hour

Exclusion Criteria:

* pregnant women,
* indication for rapid sequence induction,
* anticipation of difficult intubation,
* allergy to propofol or remifentanil,
* neurological or muscular disorder,
* combination of general anesthesia and of regional anesthesia,
* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-09; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Global score (calculated parameter which depicts the performance of the system, i.e. its capacity to maintain BIS in the desired range)

SECONDARY OUTCOMES:
consumption of propofol and remifentanil during the induction and the maintenance of the anaesthesia
number of modifications of target of propofol and remifentanil
number of episodes of hemodynamic anomalies having required a treatment
intraoperative volume loading and transfusion
extubation time, explicit memorisation
dysfunctions of each system

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch; Marc Fischler, MD, Principal Investigator — Hôpital Foch
Locations (2):
- France (2):
  - Dept of Anesthesia and Intensive Care, Hôpital Beaujon, Clichy
  - Dept of Anesthesiology, Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu N, Chazot T, Genty A, Landais A, Restoux A, McGee K, Laloe PA, Trillat B, Barvais L, Fischler M. Titration of propofol for anesthetic induction and maintenance guided by the bispectral index: closed-loop versus manual control: a prospective, randomized, multicenter study. Anesthesiology. 2006 Apr;104(4):686-95. doi: 10.1097/00000542-200604000-00012. PMID 16571963